CLINICAL TRIAL: NCT04661878
Title: Piloting a Smartphone App to Improve Treatment Adherence Among South African Adolescents Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Cape Town (Other); University of North Carolina (Other); National Institute of Mental Health (NIMH) (NIH); Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103309; K01MH118072 (NIH)
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: HIV Infections; Adolescent Behavior
Keywords: mobile health; adolescent; HIV; South Africa; social network; adherence; treatment
MeSH Terms: conditions — HIV Infections; Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MASI (Experimental): Participants randomized to the intervention condition will receive access to MASI, the smartphone app customized for this study. MASI is an adapted version of HealthMpowerment, a theory-based smartphone app with features including an anonymous interactive discussion forum, a medication and adherence tracker, a platform to ask questions to an expert, a section with engaging activities (including quizzes, self-assessments, and goal-setting activities), and a multi-media resource center.
  Interventions: Behavioral: Social Support; Behavioral: Informational Resources; Behavioral: Self-Monitoring and habit formation; Behavioral: Goal setting and action planning
- Information-only version of MASI (Active Comparator): Participants randomized to the control condition will an information-only version of MASI which will include the Resources feature and the home page.
  Interventions: Behavioral: Informational Resources

INTERVENTIONS:
Behavioral: Social Support — The app will provide opportunities for participants to interact with each other as well as trained peer mentors to receive and provide social support.
  Arms: MASI
Behavioral: Informational Resources — The app will provide opportunities for participants to review HIV-related health information in engaging formats (e.g., activities, multi-media resources, and answer to users' health questions)
Behavioral: Self-Monitoring and habit formation — The app will provide opportunities for participants to track their treatment adherence and schedule tailored reminders.
  Arms: MASI
Behavioral: Goal setting and action planning — The app will provide opportunities for participants to identify goals, select action items, and receive tailored feedback on the action plan.
  Arms: MASI

SUMMARY:
The overall goal of this pilot randomized-controlled trial (RCT) is to pilot MASI (MAsakhane Siphucule Impilo Yethu; Xhosa for "Let's empower each other and improve our health"), an ART adherence-supporting smartphone app with 50 adolescents and young adults living with HIV to assess its feasibility and acceptability and to explore preliminary effects on ART adherence and social support.

DETAILED DESCRIPTION:
Interventions that engage adolescents and young adults with HIV (AYAHIV) to improve adherence to antiretroviral therapy (ART) are urgently needed. AYAHIV repeatedly demonstrate suboptimal adherence to ART, which is associated with increased morbidity and mortality. Developing adherence-promoting interventions for AYAHIV requires an understanding of factors that shape adherence from multiple levels. Developmental theories suggest that adolescents and young adults are particularly sensitive to their social networks. Mobile health (mHealth) interventions, those that use mobile technology (e.g., smartphones apps) to transmit health information, hold promise as an effective way to improve ART adherence. These smartphone apps can be used to engage social networks and provide social support. Access to mobile phone technology is rapidly increasing among youth in South Africa, making mHealth interventions feasible and potentially scalable in this setting.

We developed MASI (MAsakhane Siphucule Impilo Yethu; Xhosa for "Let's empower each other and improve our health"), an ART adherence-supporting smartphone app for AYAHIV in South Africa. MASI was culturally adapted to the South African context using the evidence based HealthMpowerment platform. HealthMpowerment is a smartphone app-based intervention originally developed by Dr. Lisa Hightow-Weidman, and was developed based on the Institute of Medicine's Integrated Behavior Model with extensive input from youth. The app is designed to foster social support, offer tools for self-monitoring and habit formation, provide resources for goal setting and action planning, and present users with engaging informational resources.

This pilot randomized-controlled trial (RCT) is funded through a K01 Mentored Research Scientist Development Award. Prior to the pilot RCT, the study team developed and customized MASI through in-depth interviews and beta-testing with adolescents living with HIV in Cape Town. For the pilot RCT, participants will be randomized to either the full version of the MASI app or an information-only version of MASI control condition (1:1, with stratification by gender). Participants will be asked to engage with MASI for 6 months. All participants will complete baseline and follow-up assessments at 3- and 6-months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 15 years and <= 21 years
* Knows HIV status (Screened adolescents who do not know their HIV status will receive information on free voluntary HIV counseling and testing services)
* Living with HIV
* Has been prescribed medication to treat HIV
* Not attending school for learners with special needs (e.g., School of Skills)
* Has not repeated a grade in school more than once
* Has a smartphone that can download apps
* Feels comfortable using an app with content in English
* No plan to move outside of Cape Town in the next six months
* Has not previously participated in the MASI app testing phase of our study
* Able to successfully install the MASI app on their smartphone

Exclusion Criteria:

* Failure to meet any of the inclusion criteria
* Child dissent despite parent, legal guardian, caregiver informed consent

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta I Mulawa, PhD, Principal Investigator — Duke University
Locations (1):
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No
The data from this pilot randomized controlled trial will be shared after the publication of the main trial findings within the constraints required for the protection of confidentiality for study subjects. De-identified data will be available through individual requests directed to the Principal Investigator.

REFERENCES:
- [Derived] Mulawa MI, Hoare J, Knippler ET, Mtukushe B, Matiwane M, Muessig KE, Al-Mujtaba M, Wilkinson TH, Platt A, Egger JR, Hightow-Weidman LB. MASI, a Smartphone App to Improve Treatment Adherence Among South African Adolescents and Young Adults With HIV: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 19;12:e47137. doi: 10.2196/47137. PMID 37725409

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at antiretroviral therapy (ART) clinics in Cape Town, South Africa. Potential participants were identified from participant lists in other research studies who gave consent to be contacted for future research. Additional participants were recruited from public ART clinics linked to the tertiary teaching hospital, where all in-person study visits were conducted.
Groups:
- MASI: Participants randomized to the intervention condition received access to the full MASI app, including all its six features (i.e., Health Tracker, Forum, Ask the Expert, Activities, and Resources), and virtual access to MASI Peer Mentor support via the app. MASI is a comprehensive digital app intervention designed to promote ART adherence and foster social support using a strengths-based approach. MASI was adapted to the cultural context of South African adolescents and young adults living with HIV.
- Information-only Version of MASI: Participants randomized to the control condition received access to an information-only control app (consisting of only the Resource feature) delivered through MASI platform
Period: Overall Study
Arm/Group | MASI | Information-only Version of MASI
Started | 25 | 25
Completed | 19 | 20
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MASI | Information-only Version of MASI | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.24 (1.56) | 19.03 (1.60) | 18.63 (1.61)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Self-reported gender identity. Given options of male, female, or other (specify).
  Participants
    Gender identity: Female | 13 | 12 | 25
    Gender identity: Male | 11 | 13 | 24
    Gender identity: Other (participant response = non-binary) | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth.
  Participants
    Female | 13 | 12 | 25
    Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 25 | 50
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Adherence to ART, as measured by 30-day recall of days with missed ART doses [Median (Inter-Quartile Range); unit: Days with missed ART doses] — Adherence to antiretroviral therapy will be measured using the participant's self-reported number of days with missed ART doses in the past 30 days. "Thinking about the past month (30 days) on how many days did you miss taking your treatment? " Population: 1 MASI participant response "unknown"
  Days with missed ART doses
    number analyzed (Participants) | 24 | 25 | 49
    (all) | 2 [0.75 to 3] | 3 [1 to 4] | 2 [1 to 3]
Self-reported adherence in the past 30 days (binary) [Count of Participants; unit: Participants]
  Did not take all pills | 18 | 20 | 38
  Took all pills | 6 | 5 | 11
  Unknown | 1 | 0 | 1
Self-rating of adherence in the past 30 days [Count of Participants; unit: Participants] — Question text: "Thinking about the last 30 days, how would you rate how good a job you did with taking your ARVs (antiretroviral drugs) in the way that you are supposed to?"
  Participants
    Very poor | 1 | 0 | 1
    Poor | 1 | 0 | 1
    Fair | 3 | 6 | 9
    Good | 4 | 8 | 12
    Very good | 10 | 6 | 16
    Excellent | 6 | 5 | 11
Perceived Social Support and Social Isolation [Median (Inter-Quartile Range); unit: units on a scale] — Perceived social support was measured using an adapted version of the Medical Outcomes Study Social Support Survey (MOS-SS), which measures four domains of social support: emotional/informational support, tangible support, affectionate support, and positive social interaction. Outcome reported is sum of the 12 items. Total possible range: 12 - 48. Higher score indicates higher social support (better outcome).
  units on a scale | 29.0 [26.0 to 32.0] | 31.0 [25.0 to 34.0] | 29.0 [26.0 to 32.0]

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility: Number of Days Participants Log in to the App as Recorded by App Backend Paradata
Description: Feasibility will be measured by the number days participants log in to the app as recorded by app backend paradata
Time Frame: Months 1-3
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 25 | 25
Days | 15 [5 to 22] | 3 [2 to 9]

2. Primary Outcome: Intervention Feasibility: Number of Days Participants Log in to the App as Recorded by App Backend Paradata
Description: Feasibility will be measured by the number days participants log in to the app as recorded by app backend paradata
Time Frame: Months 4-6
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 25 | 25
Days | 2 [0 to 10] | 0 [0 to 4]

3. Primary Outcome: Intervention Feasibility: Total Time Participants Spend Using the App
Description: Feasibility will be measured by the total time, in minutes, participants spend using app as recorded by app backend paradata.
Time Frame: Months 1-3
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 25 | 25
Minutes | 58.95 [6.69 to 105.69] | 11.12 [3.58 to 35.53]

4. Primary Outcome: Intervention Feasibility: Total Time Participants Spend Using the App
Description: as for outcome 3
Time Frame: Months 4-6
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 25 | 25
Minutes | 5.67 [0.00 to 38.89] | 0.00 [0.00 to 6.89]

5. Primary Outcome: Intervention Feasibility: Number of Days Participants Log Medications Using the App as Recorded by App Backend Paradata
Description: Feasibility will be measured by the number of days participants log medications in the app as recorded by app backend paradata.
Time Frame: Months 1-3
Population: Feature not available (outcome not measurable) in information-only version of MASI
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 25 | 0
Days | 11 [1 to 25] |

6. Primary Outcome: Intervention Feasibility: Number of Days Participants Log Medications Using the App as Recorded by App Backend Paradata
Description: as for outcome 5
Time Frame: Months 4-6
Population: Feature not available (outcome not measurable) in information-only version of MASI
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 25 | 0
Days | 1 [0 to 5] |

7. Primary Outcome: Intervention Acceptability: Composite Score From Adapted System Usability Scale
Description: Acceptability will be measured by an average of participants' scores on an adapted version of the System Usability Scale (SUS), a scale giving a global view of subjective assessments of usability. Total possible range: 0 - 100. Higher score indicates higher usability and helpfulness (better outcome). Average SUS >68 (average for digital health apps) will be considered acceptable.
Time Frame: 3 months
Population: 24 intervention participants completed 3-month survey. Intervention acceptability not applicable for control participants.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 24 | 0
score on a scale | 70.0 [65.0 to 75.0] |

8. Primary Outcome: Intervention Acceptability: Composite Score From Adapted System Usability Scale
Description: as for outcome 7
Time Frame: 6 months
Population: 19 intervention participants completed 6-month survey. Intervention acceptability not applicable for control participants.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 19 | 0
score on a scale | 77.5 [70.0 to 80.0] |

9. Secondary Outcome: Adherence to ART, as Measured by 30-day Recall of Days With Missed ART Doses
Description: Adherence to antiretroviral therapy will be measured using the participant's self-reported number of days with missed ART doses in the past 30 days. "Thinking about the past month (30 days) on how many days did you miss taking your treatment? "
Time Frame: 3 months
Population: 24 intervention participants and 22 control participants completed 3-month survey
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 24 | 22
Days | 2.00 [0.00 to 3.00] | 2.50 [1.00 to 3.00]

10. Secondary Outcome: Adherence to ART, as Measured by 30-day Recall of Days With Missed ART Doses
Description: as for outcome 9
Time Frame: 6 months
Population: 19 intervention participants and 20 control participants completed 6-month survey
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 19 | 20
Days | 1.00 [0.00 to 3.00] | 2.00 [0.75 to 4.00]

11. Secondary Outcome: Perceived Social Support and Social Isolation Using Adapted Medical Outcomes Study Social Support Survey (MOS-SS)
Description: Perceived social support will be measured using an adapted version of the Medical Outcomes Study Social Support Survey (MOS-SS), which measures four domains of social support: emotional/informational support, tangible support, affectionate support, and positive social interaction. Outcome reported is sum of the 12 items. Total possible range: 12 - 48. Higher score indicates higher social support (better outcome).
Time Frame: 3 months
Population: 24 intervention participants and 22 control participants completed 3-month survey
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 24 | 22
score on a scale | 28.0 [25.8 to 33.3] | 26.5 [24.3 to 31.0]

12. Secondary Outcome: Perceived Social Support and Social Isolation Using Adapted Medical Outcomes Study Social Support Survey (MOS-SS)
Description: as for outcome 11
Time Frame: 6 months
Population: 19 intervention participants and 20 control participants completed 6-month survey
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | MASI | Information-only Version of MASI
Number analyzed (Participants) | 19 | 20
score on a scale | 29.0 [26.5 to 31.5] | 26.5 [24.0 to 29.0]

ADVERSE EVENTS:
Time Frame: Data were collected from time of enrollment to time of study completion, 6 months.
Arm/Group | MASI | Information-only Version of MASI
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT04661878/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT04661878/ICF_000.pdf